CLINICAL TRIAL: NCT07053098
Title: External Facilitation to Increase Prescribing of AUD Medications in the Psychiatric Setting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Melanie E Bennett, Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R34AA032051-01 (NIH)
Record Dates: First submitted 2025-06-30; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Alcohol-Related Disorders; Psychiatric Disorder
MeSH Terms: conditions — Alcohol-Related Disorders; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implementation Facilitation (Experimental): This Implementation Facilitation Intervention will include external facilitation, staff training, patient education, audit and feedback, and care coordination.
  Interventions: Other: Implementation Facilitation

INTERVENTIONS:
Other: Implementation Facilitation — Implementation facilitation is a multi-faceted process of enabling and supporting the adoption and integration of best practices into routine clinical care. It involves collaboration to understand a setting's challenges and barriers and working together to identify the best activities to address them. IF will incorporate External Facilitation, a problem-solving implementation strategy that builds supportive interpersonal relationships between an External Facilitator who is outside of the clinic who works with clinics and their identified internal champions to learn their unique barriers to implementation, use strategies to address these barriers, and plan for sustainability by integrating the practice into routine processes and workflows. Other implementation activities that will be used IF include staff training, patient education, audit and feedback, and care coordination.

SUMMARY:
This project will pilot test an implementation facilitation intervention to increase prescribing of medications for alcohol use disorder (MAUD) in patients with major mental illness and alcohol use disorder in three psychiatry treatment clinics.

DETAILED DESCRIPTION:
This project will pilot test an implementation facilitation intervention to increase prescribing of medications for alcohol use disorder (MAUD) in patients with major mental illness and alcohol use disorder in three psychiatry treatment clinics. Guided by the integrated Promoting Action on Research Implementation in Health Services framework, an external facilitator will work with each clinics' internal champion to (1) provide clinic level education on MAUD in non-specialty care settings, (2) provide clinic level training in using a standardized screen measure for alcohol use disorder, documenting screening results in the electronic health record, and documenting alcohol use disorder diagnosis in the electronic health record, (3) help internal champions use an audit and feedback system for weekly review of MAUD education and prescribing, (4) help internal champions do weekly care coordination for patients with major mental illness and alcohol use disorder, and (5) make educational materials on MAUD available on site to patients so they are informed about these treatment options. Internal champions and clinics will have access to consultation from a MAUD clinician expert. These activities will take place across pre-implementation and implementation phases and will be followed by a post-implementation facilitation sustainment period during which clinics and champions continue implementation on their own. Formative Evaluation activities will take place throughout; at the end of the sustainment phase, MAUD outcomes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* For prescribers: working as a prescriber, non-prescribing clinician, or administrator at one of the three participating clinics.
* For patients: has major mental illness (major depressive disorders, bipolar disorder, schizophrenia spectrum disorders, other psychotic disorders; posttraumatic stress disorder)
* For patients: has Alcohol Use Disorder and is being treated in one of the three participating clinics.

Exclusion Criteria:

* For all: age is less than 18 years old
* For all: not able to complete informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Prescribing medications for alcohol use disorder | 6 months after the end of implementation facilitation
  Change in the proportion of eligible patients prescribed a medication for alcohol use disorder in the clinic

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Bennett, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No